CLINICAL TRIAL: NCT05229250
Title: A Non-invasive Exercise Test for Evaluating Sport-related Arterial Blood Flow Limitation in the Leg: an Exploratory Study (NIRS and Cycling Power in Patients With FLIA)
Brief Title: NIRS and Exercise Intensity in Patients With FLIA
Status: Terminated | Type: Observational
Why Stopped: The hardware failed multiple times. As such we chose to terminate teh study
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, Martijn van Hooff, Principal Investigator, Maxima Medical Center
Other Study IDs: NL79767.015.21
Record Dates: First submitted 2021-11-19; First posted 2022-02-08 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Near-Infrared Spectroscopy; Iliac Artery Stenosis; Iliac Artery Disease; Iliac Artery Occlusion
Keywords: FLIA; NIRS; Endofibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: Subjects without FLIA
  Interventions: Other: Cycling test; Other: Occlusion tests; Device: NIRS during cycling; Device: CPET; Device: Echo-Doppler examination
- Patient subjects: Subjects with FLIA
  Interventions: Other: Cycling test; Other: Occlusion tests; Device: NIRS during cycling; Device: CPET; Device: Echo-Doppler examination

INTERVENTIONS:
Other: Cycling test — RAMP and MULTI-STAGE test
Other: Occlusion tests — Occlusion test before and after exercise
Device: NIRS during cycling — NIRS devices measuring oxygenation during exercise
Device: CPET — Cardiopulmonary exercise testing (heart rate, pulmonary gas exchange) during exercise
Device: Echo-Doppler examination — Peak systolic velocity and vascular stiffness measurements in the iliac-aortic tract

SUMMARY:
The research objectives of this project are to increase the understanding of pathophysiology and performance limitations related to sport-related flow limitation in the iliac artery (FLIA) using non-invasive measurement of muscle oxygenation at the working muscles of the leg and mechanical power output recorded during cycling exercise. Skeletal muscle oxygenation measured with Near-Infrared Spectroscopy (NIRS) is growing more accessible for use by coaches, teams, and individual athletes for use in performance testing. Describing how muscle oxygenation profiles in endurance athletes diagnosed with FLIA differ in comparison with healthy athletes may allow the use of this non-invasive, accessible measurement device for the screening of athletes at risk of developing FLIA.

The relevance of this work is that FLIA imposes risk of irreversible injury to the main artery of the leg in endurance athletes, limiting their ability to participate in exercise, with further consequences for health, fitness, and quality of life. Currently, the early course of this progressive condition is poorly understood, as early detection is difficult and hence appropriate treatment is often delayed. If impairment becomes severe, often more invasive (and risky) treatment is necessary. Earlier detection and monitoring of FLIA may allow for improved patient management and outcomes.

The design of this experiment will compare a patient group of trained cyclists diagnosed with FLIA, to healthy control subjects including cyclists of a similar fitness level without signs of FLIA. Both groups will perform an incremental ramp cycling test and an intermittent multi-stage cycling exercise test. Incremental ramp cycling testing is used as part of clinical diagnosis of FLIA, as well as performance (eg. VO2max) testing of healthy athletes. Multi-stage exercise protocols are also often used for performance testing of endurance athletes and allows for observation of (path)physiological responses during submaximal work stages. Outcome measures of muscle oxygenation kinetics with NIRS and cycling power will be analysed and compared between patients and healthy subjects.

DETAILED DESCRIPTION:
A professional cyclist covers approximately 25,000 km a year and flexes the hip 8,000,000 times in a year, while leg blood flow is in the range of 10-15 litres per minute. This poses a substantial hemodynamic load on the iliac artery. As a result, a proportion of endurance athletes develop a limitation in leg circulation due to arterial narrowing in this iliac artery. An early 'Lancet' study of the department of Sports Medicine of Máxima Medical Centre (MMC) found that 20% of professional cyclists were suffering from such a sport-related Flow Limitation in the Iliac Artery (FLIA) necessitating treatment. The incidence in recreational cyclists is unknown, but with 849,000 recreational cyclists in the Netherlands cycling over 3,000 km a year with an impressive 1,000,000 hip flexions, many of them travel similar distances as a professional cyclist, incurring similar risks for developing FLIA. If untreated, FLIA may have a pronounced impact on quality of life. Professional athletes may have to end their careers prematurely. In a substantial subset of cyclists, abnormalities may even lead to complete occlusion and/or thrombosis, with severe symptoms in daily life.

Clinical experience suggests that early detection and treatment leads to better outcomes. If diagnosed at a late stage, conservative management including changes in training behaviours and body position, or least-invasive surgical repair options will no longer suffice. The only options remaining would be to cease participation in the provocative activities altogether, or to undergo extensive and risky reconstructive vascular surgery. Understanding the early pathogenesis in order to improve detection is thus of paramount importance. Unfortunately, early detection is often missed due to the non-specific presentation of symptoms and the high level of specialisation required for clinical evaluation. There is a wide range of differential diagnoses that could contribute to the non-specific symptoms observed in the early stages of FLIA, including common musculoskeletal and tendinous injuries, mechanical or neurogenic pain referred from the low back or SI joint, hip acetabular labral tear, chronic exertional compartment syndrome, or fibromuscular dysplasia.8 Currently available diagnostic evaluations can have low sensitivity for an athletic population.

There is no single gold-standard evaluation for diagnosing FLIA. The current consensus suggests that the best single functional test is a provocative maximal exercise test on a cycle ergometer, followed by measuring blood pressure at the ankle and brachial arteries (ankle-brachial blood pressure index; ABI) in a competitive posture. In the rare case that the problem is unilateral, the sensitivity is 73%. If the problem is bilateral, the sensitivity is only 43%. Imaging techniques, including echo-Doppler examination, magnetic resonance angiogram (MRA), and computed tomography (CT) scan are more sensitive, but they are more expensive, less accessible, and not part of primary care evaluation, instead being typically reserved for investigation of more severe or complex presentations, and to guide surgical repair.

Near-infrared Spectroscopy (NIRS) is an innovative technique that measures relative oxygenation in the muscle, as the balance of oxygenated and deoxygenated haemoglobin and myoglobin. Impaired arterial leg circulation, such as observed in peripheral vascular disease (PVD) has been shown to produce a drop in oxygen saturation of skeletal muscle tissue relative to workload or exercise performance, and delays in reoxygenation kinetics after exercise and ischemic vascular occlusion tests (VOT). Consequently, NIRS may be able to detect alterations in oxygenation that are associated with the level of arterial insufficiency. We recently reported proof of concept studies regarding the potential diagnostic role of both power output and NIRS in patients with diagnosed sport-related FLIA.

Complaints reported in the early stages of FLIA are powerlessness and pain in the leg muscles when cycling near maximal exertion, which rapidly disappear with rest. Traditionally, incremental ramp cycling exercise to maximal exercise tolerance has been used as a provocative functional test, after which clinical outcome measures including ABI are tested. As the condition progresses however, symptoms can occur earlier during exercise at a lower intensity and take longer to resolve during recovery. Multi-stage exercise protocols are commonly used to understand metabolic responses related to submaximal exercise intensity. Therefore, a progressive multi-stage cycling protocol with brief recovery intervals between work intervals will be introduced. This protocol is designed to allow for multiple opportunities to evaluate work and recovery responses in an intensity-dependent manner. Subjective symptoms, performance impairments (including limitations to cycling power output) and muscle oxygenation kinetic delays will be evaluated across submaximal workloads including after maximal intensity.

Understanding the onset of symptoms and objective signs of flow limitation with progressive exercise intensity will improve understanding of severity and progression of this condition. These outcome measures will be compared to healthy subjects, in order to develop normative values related to healthy performance, compared to pathological impairment. The use of a common multi-stage performance assessment protocol will improve the applicability of using this approach for screening and early detection of FLIA outside of a specialised vascular clinic.

It has been suggested that altered vascular function and structure may contribute to the appearance of symptoms in patients in which obvious stenosis or intraluminal disease is not apparent on imaging. In addition to standard clinical evaluation of the aortoiliac tract with echo-Doppler ultrasound, vascular flow velocity will be recorded for later offline analysis of pulse wave velocity as a measurement of arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years and ≤ 40 years
* Trained cyclist or triathlete regularly training at least ~3/week for at least five years and identifying with a particular cycle-sport

Exclusion Criteria:

* Earlier vascular iliac surgery
* Microvascular abnormalities (e.g. diabetes),
* Vascular abnormalities outside of the iliac region,
* Heart failure (New York Heart Association class >I),
* Orthopedic/neurological entities potentially limiting exercise capacity,
* Obesity.
* Adipose tissue thickness > 7.5 mm

These excluding conditions are considered as medical safety precautions to maximal exercise or as risk of unexpected pathophysiological effects confounding our primary outcome measures.

It is known that a high level of adipose tissue thickness (ATT) influences the accuracy of NIRS measurement of underlying muscular tissue. A > 7.5 mm ATT cut-off point at the site of NIRS measurement determined with a skinfold caliper (Harpenden, Baty International West Sussex, UK) was chosen. The ATT is calculated as half the skinfold thickness.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited after the diagnosis of FLIA is given during weekly standard clinical care.
  Healthy subjects will be recruited from local cycling clubs. They completed a standardized questionnaire excluding presence of risk factors such as smoking and positive cardiovascular family history. Candidates with FLIA were excluded. Candidates who fulfilled all study criteria, served as the control group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Power-deoxygenation (PD) profile | During cyclingtest day 1
  Power-deoxygenation (PD) profile: The ratio of power output to deoxygenation (eg. power/deoxy[heme]) as a proxy for the metabolic disturbance at the working muscle relative to the workload.
Near Infrared Spectroscopy (NIRS) deoxygenation parameters | During cyclingtest day 1
  Baseline: Average 60-second value before the start of exercise. min: the minimum 5-second mean value attained during exercise. max: the maximum 5-second mean value attained typically during the recovery after exercise.
  Δexercise amplitude: the difference between baseline and minimum values.
Near Infrared Spectroscopy (NIRS) deoxygenation parameters | During cyclingtest day 2
  Baseline: Average 60-second value before the start of exercise. min: the minimum 5-second mean value attained during exercise. max: the maximum 5-second mean value attained typically during the recovery after exercise.
  Δexercise amplitude: the difference between baseline and minimum values.
NIRS delta_recovery amplitude | During cyclingtest day 1
  The difference between minimum and maximum value.
NIRS delta_recovery amplitude | During cyclingtest day 2
  The difference between minimum and maximum value.
NIRS reoxygenation kinetics: tau | Immediately after exercise day 1
  Time constant (tau, in seconds): the time constant parameter of a monoexponential curve fit to the reoxygenation profile after each work stage.
NIRS reoxygenation kinetics: Time delay | Immediately after exercise day 1
  Time delay (TD, in seconds): the delay before systematic rise in oxygenation after each work stage.
NIRS reoxygenation kinetics: Mean Response Time | Immediately after exercise day 1
  Mean response time (MRT, in seconds): the sum of TD and tau.
NIRS reoxygenation kinetics: Half value time | Immediately after exercise day 1
  Half value recovery time (HVT, in seconds): the time required to reoxygenate half of the total amplitude during recovery after each work stage.
NIRS reoxygenation kinetics: Peak reoxygenation rate | Immediately after exercise day 1
  Peak reoxygenation rate (SmO2/sec): a linear estimation of the peak resaturation slope, representing the magnitude of greatest mismatch between oxygen supply and utilization at the tissue during recovery kinetics, after each work stage.
NIRS reoxygenation kinetics: Peak reoxygenation MRT | Immediately after exercise day 1
  Peak reoxygenation MRT: an estimate of the time to occurrence of the peak reoxygenation rate, analogous to the MRT in a monoexponential curve, and representing the balance of recovery kinetics of oxygen supply and utilization in the tissue after each work stage.
NIRS reoxygenation kinetics: tau | Immediately after exercise day 2
  Time constant (tau, in seconds): the time constant parameter of a monoexponential curve fit to the reoxygenation profile after each work stage.
NIRS reoxygenation kinetics: Time delay | Immediately after exercise day 2
  Time delay (TD, in seconds): the delay before systematic rise in oxygenation after each work stage.
NIRS reoxygenation kinetics: Mean response time | Immediately after exercise day 2
  Mean response time (MRT, in seconds): the sum of TD and tau.
NIRS reoxygenation kinetics: Half Value time | Immediately after exercise day 2
  Half value recovery time (HVT, in seconds): the time required to reoxygenate half of the total amplitude during recovery after each work stage.
NIRS reoxygenation kinetics: Peak reoxygenation rate | Immediately after exercise day 2
  Peak reoxygenation rate (SmO2/sec): a linear estimation of the peak resaturation slope, representing the magnitude of greatest mismatch between oxygen supply and utilization at the tissue during recovery kinetics, after each work stage.
NIRS reoxygenation kinetics: Peak reoxygenation MRT | Immediately after exercise day 2
  Peak reoxygenation MRT: an estimate of the time to occurrence of the peak reoxygenation rate, analogous to the MRT in a monoexponential curve, and representing the balance of recovery kinetics of oxygen supply and utilization in the tissue after each work stage.

SECONDARY OUTCOMES:
Recovery kinetics VO2/NIRS comparison | After stages/maximal exercise. This is an offline analyses and therefore takes the time of the stage (1 minute for in between blocks; 5 minutes for maximal exercise)
  To describe skeletal muscle oxygenation kinetics vs pulmonary oxygen uptake kinetics in both healthy cyclists and patients with FLIA
Vascular Occlusion Test - Reactive Hyperemia Area Under The Curve | Before cycling test day 1
  Reactive Hyperemia area under the curve: the area of the NIRS signal (eg. SmO2⋅sec) will be calculated during the recovery from occlusion, as the total area under the curve and above the baseline value before cuff inflation during the first 4-minutes of recovery.
  (This will be calculated from the same VOT for Outcome 1
Multiple reoxygenation kinetics - Primary Component Time constant tau | Between intervention day 1 (1-minute stages of block-protocol) and immediately after the intervention day 2 (ramp maximal test)
  Primary component time constant (tau): the time constant parameter of a monoexponential curve fit to the rise in VO2 at the start of each work stage.
Multiple reoxygenation kinetics - Cardiodynamic component time delay | Between intervention day 1 (1 minustages of block-protocol) and immediately after the intervention day 2 (ramp maximal test)
  Cardiodynamic component time delay (TD): the delay before systematic rise in VO2 at the start of each work stage.
Multiple reoxygenation kinetics - Δdeoxy[heme] / ΔVO2 onset kinetics | During intervention day 1 (stages of block-protocol)
  Δdeoxy[heme] / ΔVO2 onset kinetics: The oxygenation and VO2 curves will be normalized at the start of each work stage to a starting baseline and the eventual steady-state, as 0-100% of the response profile. The relative overshoot of Δdeoxy[heme] vs ΔVO2 can then be used to describe the matching of perfusive O2 delivery to O2 extraction.
Multiple reoxygenation kinetics - Δdeoxy[heme] / ΔVO2 recovery kinetics | Between intervention day 1 (stages of block-protocol) and immediately after the intervention day 2 (ramp maximal test)
  Δdeoxy[heme] / ΔVO2 recovery kinetics: The same comparison of the response profiles of deoxy[heme] and VO2 will be performed during recovery after work stages.
Vascular Occlusion Test (VOT): Microvascular Responsiveness | Before and after cycling test day 1
  Microvascular Responsiveness (peak reoxygenation rate, eg. SmO2/sec): the linear slope of reoxygenation when the occlusion cuff is removed will be taken as the rate of reperfusion, representing microvascular responsiveness, a proxy for vasodilatory capacity and vascular function.
Vascular Occlusion Test (VOT): Reactive Hyperemia | Before and after cycling test day 1
  Reactive Hyperemia area under the curve: the area of the NIRS signal (eg. SmO2⋅sec) will be calculated during the recovery from occlusion, as the total area under the curve and above the baseline value before cuff inflation during the first 4-minutes of recovery.
  Calculated from same in VOT (Outcome 7)
Clinical Assessment | During the same examination-appointment. The PSV will be measured following measurments of the arterial stiffness. This takes about 10 minutes for both sides.
  Peak systolic velocity (PSV): Measurement of PSV at the external iliac artery with echo-Doppler ultrasound, before and after exercise, and with and without provocative maneuvers can be discriminative for FLIA.
Clinical Assessment | Immediately after maximal exercise day 1
  Ankle brachial index (ABI): Blood pressures will be taken at bilateral ankles and from the arm both before and after exercise. The ratio of ankle and brachial pressures adjusted for height, and a bilateral difference can be discriminative for FLIA.
Clinical Assessment | Immediately after maximal exercise day 2
  Ankle brachial index (ABI): Blood pressures will be taken at bilateral ankles and from the arm both before and after exercise. The ratio of ankle and brachial pressures adjusted for height, and a bilateral difference can be discriminative for FLIA.
Clinical Assessment | Before exercise day 1, the arterial stiffness will be measured by the vascular technician. While this will be analyzed offline, this takes a few minutes.
  Arterial stiffness with echo-Doppler: Arterial pulse wave velocities will be measured at the carotid and external iliac/femoral arteries with echo-Doppler ultrasound, before and after exercise. The velocity of propagation of the pulse wave is taken as an index of arterial stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: M van Hooff, MSc, Principal Investigator — Maxima Medical Center
Locations (1):
- Maxima MC, Veldhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Hooff M, Schep G, Bender M, Scheltinga M, Savelberg H. Sport-related femoral artery occlusion detected by near-infrared spectroscopy and pedal power measurements: a case report. Phys Sportsmed. 2021 May;49(2):241-244. doi: 10.1080/00913847.2020.1796182. Epub 2020 Jul 26. PMID 32713244
- [Background] van Hooff M, Schep G, Meijer E, Bender M, Savelberg H. Near-Infrared Spectroscopy Is Promising to Detect Iliac Artery Flow Limitations in Athletes: A Pilot Study. J Sports Med (Hindawi Publ Corp). 2018 Dec 20;2018:8965858. doi: 10.1155/2018/8965858. eCollection 2018. PMID 30671480
- [Background] Schep G, Bender MH, van de Tempel G, Wijn PF, de Vries WR, Eikelboom BC. Detection and treatment of claudication due to functional iliac obstruction in top endurance athletes: a prospective study. Lancet. 2002 Feb 9;359(9305):466-73. doi: 10.1016/s0140-6736(02)07675-4. PMID 11853791
- [Background] Bender MH, Schep G, de Vries WR, Hoogeveen AR, Wijn PF. Sports-related flow limitations in the iliac arteries in endurance athletes: aetiology, diagnosis, treatment and future developments. Sports Med. 2004;34(7):427-42. doi: 10.2165/00007256-200434070-00002. PMID 15233596
- [Background] Peach G, Schep G, Palfreeman R, Beard JD, Thompson MM, Hinchliffe RJ. Endofibrosis and kinking of the iliac arteries in athletes: a systematic review. Eur J Vasc Endovasc Surg. 2012 Feb;43(2):208-17. doi: 10.1016/j.ejvs.2011.11.019. Epub 2011 Dec 19. PMID 22186674
- [Background] Hinchliffe RJ. Iliac Artery Endofibrosis. Eur J Vasc Endovasc Surg. 2016 Jul;52(1):1-2. doi: 10.1016/j.ejvs.2016.04.006. Epub 2016 May 6. No abstract available. PMID 27161328
- [Background] INSITE Collaborators (INternational Study group for Identification and Treatment of Endofibrosis). Diagnosis and Management of Iliac Artery Endofibrosis: Results of a Delphi Consensus Study. Eur J Vasc Endovasc Surg. 2016 Jul;52(1):90-8. doi: 10.1016/j.ejvs.2016.04.004. Epub 2016 May 17. PMID 27209899
- [Background] Khan A, Al-Dawoud M, Salaman R, Al-Khaffaf H. Management of Endurance Athletes with Flow Limitation in the Iliac Arteries: A Case Series. EJVES Short Rep. 2018 Jul 20;40:7-11. doi: 10.1016/j.ejvssr.2018.06.001. eCollection 2018. PMID 30101198
- [Background] Peake LK, D'Abate F, Farrah J, Morgan M, Hinchliffe RJ. The Investigation and Management of Iliac Artery Endofibrosis: Lessons Learned from a Case Series. Eur J Vasc Endovasc Surg. 2018 Apr;55(4):577-583. doi: 10.1016/j.ejvs.2018.01.018. Epub 2018 Mar 13. PMID 29548540
- [Background] Schep G, Bender MH, Schmikli SL, Mosterd WL, Hammacher ER, Scheltinga M, Wijn PF. Recognising vascular causes of leg complaints in endurance athletes. Part 2: the value of patient history, physical examination, cycling exercise test and echo-Doppler examination. Int J Sports Med. 2002 Jul;23(5):322-8. doi: 10.1055/s-2002-33142. PMID 12165882
- [Background] Barstow TJ. Understanding near infrared spectroscopy and its application to skeletal muscle research. J Appl Physiol (1985). 2019 May 1;126(5):1360-1376. doi: 10.1152/japplphysiol.00166.2018. Epub 2019 Mar 7. PMID 30844336
- [Background] Perrey S, Ferrari M. Muscle Oximetry in Sports Science: A Systematic Review. Sports Med. 2018 Mar;48(3):597-616. doi: 10.1007/s40279-017-0820-1. PMID 29177977
- [Background] Boezeman RP, Moll FL, Unlu C, de Vries JP. Systematic review of clinical applications of monitoring muscle tissue oxygenation with near-infrared spectroscopy in vascular disease. Microvasc Res. 2016 Mar;104:11-22. doi: 10.1016/j.mvr.2015.11.004. Epub 2015 Nov 11. PMID 26576829
- [Background] Cornelis N, Chatzinikolaou P, Buys R, Fourneau I, Claes J, Cornelissen V. The Use of Near Infrared Spectroscopy to Evaluate the Effect of Exercise on Peripheral Muscle Oxygenation in Patients with Lower Extremity Artery Disease: A Systematic Review. Eur J Vasc Endovasc Surg. 2021 May;61(5):837-847. doi: 10.1016/j.ejvs.2021.02.008. Epub 2021 Mar 30. PMID 33810977
- [Background] Kleinloog JPD, van Hooff M, Savelberg HHCM, Meijer EJ, Schep G. Pedal power measurement as a diagnostic tool for functional vascular problems. Clin Biomech (Bristol). 2019 Jan;61:211-216. doi: 10.1016/j.clinbiomech.2018.12.020. Epub 2018 Dec 21. PMID 30597482
- [Background] Arnold J, Yogev A, Koehle MS. Evaluating Arterial Blood Flow Limitation Using Muscle Oxygenation and Cycling Power. Clin J Sport Med. 2022 May 1;32(3):e268-e275. doi: 10.1097/JSM.0000000000000942. Epub 2021 May 7. PMID 34009787
- [Background] Jamnick NA, Botella J, Pyne DB, Bishop DJ. Manipulating graded exercise test variables affects the validity of the lactate threshold and V ⁢ O 2 ⁢ peak . PLoS One. 2018 Jul 30;13(7):e0199794. doi: 10.1371/journal.pone.0199794. eCollection 2018. PMID 30059543
- [Background] Ihsan M, Abbiss CR, Lipski M, Buchheit M, Watson G. Muscle oxygenation and blood volume reliability during continuous and intermittent running. Int J Sports Med. 2013 Jul;34(7):637-45. doi: 10.1055/s-0032-1331771. Epub 2013 Mar 22. PMID 23526593
- [Background] Skovereng K, Ettema G, van Beekvelt M. Local muscle oxygen consumption related to external and joint specific power. Hum Mov Sci. 2016 Feb;45:161-71. doi: 10.1016/j.humov.2015.11.009. Epub 2015 Dec 1. PMID 26650852
- [Background] Heres HM, Schoots T, Tchang BCY, Rutten MCM, Kemps HMC, van de Vosse FN, Lopata RGP. Perfusion dynamics assessment with Power Doppler ultrasound in skeletal muscle during maximal and submaximal cycling exercise. Eur J Appl Physiol. 2018 Jun;118(6):1209-1219. doi: 10.1007/s00421-018-3850-y. Epub 2018 Mar 22. PMID 29569054
- [Background] Bopp CM, Townsend DK, Barstow TJ. Characterizing near-infrared spectroscopy responses to forearm post-occlusive reactive hyperemia in healthy subjects. Eur J Appl Physiol. 2011 Nov;111(11):2753-61. doi: 10.1007/s00421-011-1898-z. Epub 2011 Mar 16. PMID 21409404
- [Background] Niemeijer VM, Spee RF, Jansen JP, Buskermolen AB, van Dijk T, Wijn PF, Kemps HM. Test-retest reliability of skeletal muscle oxygenation measurements during submaximal cycling exercise in patients with chronic heart failure. Clin Physiol Funct Imaging. 2017 Jan;37(1):68-78. doi: 10.1111/cpf.12269. Epub 2015 Jul 3. PMID 26147875
- [Background] Chirinos JA, Segers P, Hughes T, Townsend R. Large-Artery Stiffness in Health and Disease: JACC State-of-the-Art Review. J Am Coll Cardiol. 2019 Sep 3;74(9):1237-1263. doi: 10.1016/j.jacc.2019.07.012. PMID 31466622
- [Background] Stocker F, Von Oldershausen C, Paternoster FK, Schulz T, Oberhoffer R. End-exercise DeltaHHb/DeltaVO2 and post-exercise local oxygen availability in relation to exercise intensity. Clin Physiol Funct Imaging. 2017 Jul;37(4):384-393. doi: 10.1111/cpf.12314. Epub 2015 Nov 17. PMID 26576503
- [Background] Rosenberry R, Nelson MD. Reactive hyperemia: a review of methods, mechanisms, and considerations. Am J Physiol Regul Integr Comp Physiol. 2020 Mar 1;318(3):R605-R618. doi: 10.1152/ajpregu.00339.2019. Epub 2020 Feb 5. PMID 32022580
- [Background] McLay KM, Fontana FY, Nederveen JP, Guida FF, Paterson DH, Pogliaghi S, Murias JM. Vascular responsiveness determined by near-infrared spectroscopy measures of oxygen saturation. Exp Physiol. 2016 Jan;101(1):34-40. doi: 10.1113/EP085406. Epub 2015 Dec 6. PMID 26498127